CLINICAL TRIAL: NCT02408120
Title: Benefits of Insulin Supplementation for Correction of Hyperglycemia in Patients With Type 2 Diabetes Treated With Basal Bolus Insulin Regimen
Brief Title: Benefits of Insulin Supplementation for Correction of Hyperglycemia in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Priyathama Vellanki, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00078695
Record Dates: First submitted 2015-03-27; First posted 2015-04-03 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Hyperglycemia; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Hypoglycemia | interventions — Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Aspart for BG > 140 mg/dL (Active Comparator): Subjects will consist of hospitalized patients with type 2 diabetes and be randomized to receive insulin glargine once daily and insulin aspart divided in three equal doses before meals. Supplemental insulin aspart will be given before meals and at bedtime to subjects with blood glucose (BG) levels >140 mg/dL.
  Interventions: Drug: Insulin glargine; Drug: Insulin aspart; Drug: Supplemental insulin aspart
- Insulin Aspart for BG > 260 mg/dL (Active Comparator): Subjects will consist of hospitalized patients with type 2 diabetes and be randomized to receive insulin glargine once daily and insulin aspart divided in three equal doses before meals. Supplemental insulin aspart will be given before meals and at bedtime to subjects with blood glucose (BG) levels >260 mg/dL.
  Interventions: Drug: Insulin glargine; Drug: Insulin aspart; Drug: Supplemental insulin aspart

INTERVENTIONS:
Drug: Insulin glargine — Half of total daily dose (TDD) will be given as insulin glargine and will be given once daily, at the same time of the day.
  Daily insulin dose will be adjusted as follow:
  * If the fasting and pre-dinner BG is between 100 - 140 mg/dL in the absence of hypoglycemia the previous day: no change
  * If the fasting and pre-dinner BG is between 140 - 180 mg/dL in the absence of hypoglycemia: increase basal insulin by 10% every day
  * If the fasting and pre-dinner BG is >180 mg/dL in the absence of hypoglycemia the previous day: increase basal insulin dose by 20% every day
  * If the fasting and pre-dinner BG is between 70 - 99 mg/dL in the absence of hypoglycemia: decrease TDD (basal and prandial) insulin dose by 10% every day
  * If a patient develops hypoglycemia (BG <70 mg/dL), the insulin TDD (basal and prandial) should be decreased by 20%.
  Other Names: Lantus (glargine)
Drug: Insulin aspart — Half of total daily dose will be given as insulin aspart and in three equally divided doses before each meal. To prevent hypoglycemia, if a subject is not able to eat, the dose of aspart will be held.
  Daily insulin dose will be adjusted as follow:
  * If the fasting and pre-dinner BG is between 100 - 140 mg/dL in the absence of hypoglycemia the previous day: no change
  * If the fasting and pre-dinner BG is between 140 - 180 mg/dL in the absence of hypoglycemia: increase basal insulin by 10% every day
  * If the fasting and pre-dinner BG is >180 mg/dL in the absence of hypoglycemia the previous day: increase basal insulin dose by 20% every day
  * If the fasting and pre-dinner BG is between 70 - 99 mg/dL in the absence of hypoglycemia: decrease TDD (basal and prandial) insulin dose by 10% every day
  * If a patient develops hypoglycemia (BG <70 mg/dL), the insulin TDD (basal and prandial) should be decreased by 20%.
  Other Names: Novolog
Drug: Supplemental insulin aspart — Insulin aspart will be administered following the supplemental insulin scale protocol.
  For the arm receiving supplemental insulin aspart at BG levels greater than 140 mg/dL, then supplemental insulin scale is as follows:
  * BG >141-180 mg/dL; 2-4 units of insulin aspart
  * BG between 181-220 mg/dL; 3-6 units of insulin aspart
  * BG between 221-260 mg/dL; 4-8 units of insulin aspart
  * BG between 261-300 mg/dL; 5-10 units of insulin aspart
  * BG between 301-350 mg/dL; 6-12 units of insulin aspart
  * BG between 351-400 mg/dL; 7-14 units of insulin aspart
  * BG > 400 mg/dL; 8-16 units of insulin aspart
  For the arm receiving supplemental insulin aspart at BG levels greater than 260 mg/dL, then supplemental insulin scale is as follows:
  * BG between 261-300 mg/dL; 5-10 units of insulin aspart
  * BG between 301-350 mg/dL; 6-12 units of insulin aspart
  * BG between 351-400 mg/dL; 7-14 units of insulin aspart
  * BG > 400 mg/dL; 8-16 units of insulin aspart
  Other Names: Novolog

SUMMARY:
The purpose of this study is to test whether using extra doses of aspart insulin to correct blood sugars before meals improves the care of patients with type 2 diabetes in the hospital who are already receiving the standard of care treatment with glargine and aspart insulin injections to control blood sugar levels. Studies done in the past indicate that blood sugar levels are controlled on the standard treatment of insulin and that most patients do not need the small extra dose of insulin at bedtime. The investigators want to test if there is any benefit to giving patients extra doses of insulin during the day to correct the high blood sugars.

DETAILED DESCRIPTION:
The management of patients with Type 2 diabetes involves treatment with two different types of insulin injections to control blood sugar levels. The doses of the two types of insulins, glargine insulin and aspart insulin are adjusted daily through the hospital stay based on blood sugar levels. Many times, in addition to glargine and aspart insulin at meals, additional small doses of aspart insulin are given to correct high blood sugar levels. It has not been determined if using these extra doses of aspart insulin to correct blood sugars before meals improves care of the patients. Studies done in the past indicate that blood sugar levels are well controlled on the standard treatment of the two insulins and that most patients do not need the small extra dose of insulin at bedtime. This study will test if insulin supplementation improves glycemic control and prevents hypoglycemia in insulin treated patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects admitted to the hospital with acute or chronic medical illnesses or for elective and emergency surgical illness or trauma
2. Known history of Type 2 diabetes mellitus for >3 months
3. Treated with either diet alone, any combination of oral antidiabetic agents, non-insulin injectables or insulin therapy
4. Blood glucose levels between >140 mg and <400 mg/dL without laboratory evidence of diabetic ketoacidosis

Exclusion Criteria:

1. Hyperglycemia without a history of diabetes
2. Subjects with acute critical illness admitted to the ICU or expected to require ICU admission
3. Subjects receiving continuous insulin infusion
4. Clinically relevant hepatic disease
5. Corticosteroid therapy
6. Serum creatinine ≥ 3.5 mg/dL and/or glomerular filtration rate (GFR) <30
7. Subjects unable to sign consent
8. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2015-10; Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priyathama Vellanki, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vellanki P, Cardona S, Galindo RJ, Urrutia MA, Pasquel FJ, Davis GM, Fayfman M, Migdal A, Peng L, Umpierrez GE. Efficacy and Safety of Intensive Versus Nonintensive Supplemental Insulin With a Basal-Bolus Insulin Regimen in Hospitalized Patients With Type 2 Diabetes: A Randomized Clinical Study. Diabetes Care. 2022 Oct 1;45(10):2217-2223. doi: 10.2337/dc21-1606. PMID 35675498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 226 subjects consented from October 2015 to December 2019. Two subjects withdrew or left the hospital prior to randomization.
Period: Overall Study
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Started | 112 | 112
Completed | 108 | 107
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Treatment Refusal | 1 | 0
Not completed — Received Steroids | 1 | 1
Not completed — Discharged same day | 1 | 1
Not completed — Did not receive insulin | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL | Total
Number analyzed (Participants) | 108 | 107 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 78 | 154
  >=65 years | 32 | 29 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 115
  Male | 51 | 49 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 92 | 82 | 174
  White | 15 | 22 | 37
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 108 | 107 | 215

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily BG Levels
Description: Blood glucose (BG) will be measured, and mean daily BG levels will be calculated.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
mg/dL | 172 (38.2) | 173 (43)

2. Secondary Outcome: Mean Blood Glucose Levels Before Lunch
Description: The blood glucose levels will be assessed prior to lunch using a glucose meter.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
mg/dL | 160 (16) | 172 (14)

3. Secondary Outcome: Mean Blood Glucose Levels at Bedtime
Description: The blood glucose levels will be assessed at bedtime using a glucose meter.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
mg/dl | 157 (18) | 171 (9)

4. Secondary Outcome: Mean Blood Glucose Levels Before Dinner
Description: The blood glucose levels will be assessed before dinner using a glucose meter.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
mg/dL | 151 (19) | 160 (10)

5. Secondary Outcome: Number of Hypoglycemia Events
Description: The number of occurrences of hypoglycemia (blood glucose levels < 70 mg/dL) will be recorded.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Number; unit: number of events
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
number of events | 16 | 15

6. Secondary Outcome: Incidence of Hyperglycemia
Description: The number of occurrences of hyperglycemia (blood glucose levels > 260 mg/dL) will be recorded.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Number; unit: number of events
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
number of events | 45 | 42

7. Secondary Outcome: Number of Blood Glucose Readings Within 100-140 mg/dL Range
Description: The number of blood glucose readings that are in the target range of 100-140 mg/dL will be recorded.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Number; unit: number of readings
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
number of readings | 59 | 57

8. Secondary Outcome: Average Number of Days of Hospital Stay
Description: The average number of days in the hospital for subjects will be calculated.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
days | 4 [3 to 7.5] | 4 [3 to 9]

9. Secondary Outcome: Mortality
Description: The total number of subject deaths during hospital stay will be recorded.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
Participants | 1 | 0

10. Secondary Outcome: Number of Subjects That Experienced Hospital Complications
Description: The total number of subjects in which hospital complications occurred prior to discharge will be recorded. These complications will mainly be cases of nosocomial infections, pneumonia, bacteremia, respiratory failure, and acute kidney injury [rise of serum creatinine >0.5 mg/dL (or 50%) of baseline value]. Nosocomial infections will be diagnosed based on standardized Centers for Disease Control (CDC) criteria.
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
Participants | 11 | 12

11. Secondary Outcome: Mean Daily Dose of Insulin
Description: Daily dose of insulin will be recorded
Time Frame: 5 days (average time of discharge from the hospital)
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
Number analyzed (Participants) | 108 | 107
units/day | 47 (43) | 41 (30)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Insulin Aspart for BG > 140 mg/dL | Insulin Aspart for BG > 260 mg/dL
All-Cause Mortality (participants affected / at risk) | 1/108 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/107
Other Adverse Events (participants affected / at risk) | 11/108 | 12/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Aspart for BG > 140 mg/dL (N=108) | Insulin Aspart for BG > 260 mg/dL (N=107)
Acute Kidney Injury (Renal and urinary disorders) | 10 | 11
Infection (Infections and infestations) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT02408120/Prot_SAP_000.pdf